CLINICAL TRIAL: NCT04762576
Title: Diagnosis and Management of Impaired Thrombin Generation in Cardiac Surgery
Brief Title: Thrombin in Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: 20-5726
Record Dates: First submitted 2021-02-02; First posted 2021-02-21 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Thrombin; Hemostatic Disorder; Surgical Blood Loss; Coagulation Disorder; Cardiovascular Surgical Procedures
MeSH Terms: conditions — Hemostatic Disorders; Blood Loss, Surgical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples will be retained for CAT analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiac Surgical Patients: All consenting adults undergoing cardiac surgery at Toronto General Hospital.

SUMMARY:
Coagulopathy, bleeding, and transfusion are common in cardiac surgical patients. Our collaborator has developed a novel point of care device that can be used to assess thrombin generation in real-time in cardiac surgical patients. The investigators will measure thrombin generation using our novel device and compare it to standard methods, while examining the association of thrombin parameters with bleeding and other clinical outcomes.

DETAILED DESCRIPTION:
This is a prospective observational cohort study of 200 cardiac surgical patients. Thrombin generation via our novel point of care thrombin generation assay as well as calibrated automated thrombography (CAT) will be measured at three time points: (1) before surgery; (2) post-CPB after heparin reversal with protamine; (3) at the time of chest closure or 60 minutes after heparin reversal with protamine. Clinicians will remain blinded to the measures. Recruitment will continue until the investigators enroll 50 patients with significant impaired thrombin generation capacity (>50% drop from baseline) and 50 patients who receive hemostatic therapies. Patients will be followed for 7 days postoperatively to assess individual products transfused.

ELIGIBILITY:
Inclusion Criteria:

-All adult patients (> 18 years of age) undergoing cardiac surgery at Toronto General Hospital will be offered participation.

Exclusion Criteria:

-Patients who are unable to consent to the study or who refuse participation will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cardiovascular disease undergoing cardiac surgical procedures at Toronto General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Thrombin Generation, as assessed by the Endogenous Thrombin Potential (ETP) | The change in thrombin generation will be assessed from preoperative baseline up until 12 hours post-operatively
  The primary thrombin generation parameter of interest is the endogenous thrombin potential, or ETP, expressed in nM*min. The change in thrombin generation in patients undergoing cardiac surgery before and after cardiopulmonary bypass using our new point-of-care thrombin sensor and the established laboratory-based calibrated automated thrombogram (CAT) assay will be assessed.
Thrombin Generation, as assessed by the Lag Time | The change in thrombin generation will be assessed from preoperative baseline up until 12 hours post-operatively
  The co-primary thrombin generation parameter of interest is the Lag Time, expressed in seconds. The change in thrombin generation in patients undergoing cardiac surgery before and after cardiopulmonary bypass using our new point-of-care thrombin sensor and the established laboratory-based calibrated automated thrombogram (CAT) assay will be assessed.
Thrombin Generation, as assessed by the Time to Peak | The change in thrombin generation will be assessed from preoperative baseline up until 12 hours post-operatively
  The co-primary thrombin generation parameter of interest is the Time to Peak, expressed in seconds. The change in thrombin generation in patients undergoing cardiac surgery before and after cardiopulmonary bypass using our new point-of-care thrombin sensor and the established laboratory-based calibrated automated thrombogram (CAT) assay will be assessed.
Thrombin Generation, as assessed by the Peak Height | The change in thrombin generation will be assessed from preoperative baseline up until 12 hours post-operatively
  The co-primary thrombin generation parameter of interest is the Peak Height, expressed in nM. The change in thrombin generation in patients undergoing cardiac surgery before and after cardiopulmonary bypass using our new point-of-care thrombin sensor and the established laboratory-based calibrated automated thrombogram (CAT) assay will be assessed.

SECONDARY OUTCOMES:
Total Units of Red Blood Cells Transfused | From intra-operatively up to 12 hours post-operatively
  The total number of red blood cells units transfused will be recorded
Total Units of Platelets Transfused | From intra-operatively up to 12 hours post-operatively
  The total number of platelets units transfused will be recorded
Total Units of Frozen Plasma Transfused | From intra-operatively up to 12 hours post-operatively
  The total number of frozen plasma units transfused will be recorded
Total amount of Prothrombin Complex Concentrates transfused | From intra-operatively up to 12 hours post-operatively
  The total number of prothrombin complex concentrate units will be recorded
Total amount of Fibrinogen Concentrate transfused | From intra-operatively up to 12 hours post-operatively
  The total number of grams of fibrinogen concentrate transfused will be recorded

OTHER OUTCOMES:
Chest tube drainage | From intra-operatively to within 12 hours post-operatively
  Blood loss from chest tube drainage will be assessed in mL
Return to the Operating Room for Bleeding or Delayed Chest Closure | From intra-operatively to within 12 hours post-operatively
  Instances of return to the operating room for re-exploration or a delay in chest closure will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Bartoszko, MD MSc FRCPC, Principal Investigator — Toronto General Hospital - University Health Network; Keyvan Karkouti, MD MSc FRCPC, Principal Investigator — Toronto General Hospital - University Health Network
Locations (1):
- Toronto General Hospital - University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No